CLINICAL TRIAL: NCT05107453
Title: Serratus Anterior Plane Block for Minimal Invasive Cardiac Surgery: a Single Center Randomized-controlled Trial
Brief Title: Serratus Anterior Plane Block for Minimal Invasive Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Bart Vaes, MD, Principal Investigator, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MMS.2021.042
Record Dates: First submitted 2021-10-28; First posted 2021-11-04 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Minimal Invasive Cardiac Surgery; Mitral Valve Surgery; Aortic Valve Replacement; Minimal Invasive Direct Coronary Artery Bypass
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patient, intensivist, ICU nurses and data manager are blinded for the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAPB (Active Comparator): The IMP is levobupivacaine 0,25%, 2,5 mg/ml, solution for injection. The dosage scheme is as following:1.25 mg/kg levobupivacaine 0,25%, with a maximum of 100 mg, As the standard anaesthetic management already contains levobupivacaine, a maximum dosage of 100 mg (40 ml) levobupivacaine will be administered during the SAPB.
  The IMP is given via ultrasound-guided infiltration, in plane, midaxillary, 4-5th rib, between the latissimus dorsi and serratus anterior muscle, at the end of surgery.
  Interventions: Drug: Levobupivacaine
- Control (No Intervention)

INTERVENTIONS:
Drug: Levobupivacaine — The Investigational Medical Product (IMP) is levobupivacaine 0,25%, 2,5 mg/ml, solution for injection. The dosage scheme is as following:1.25 mg/kg levobupivacaine 0,25%, with a maximum of 100 mg, As the standard anaesthetic management already contains levobupivacaine, a maximum dosage of 100 mg (40 ml) levobupivacaine will be administered during the SAPB.
  The IMP is given via ultrasound-guided infiltration, in plane, midaxillary, 4-5th rib, between the latissimus dorsi and serratus anterior muscle, at the end of surgery.
  Arms: SAPB

SUMMARY:
Analgesia in cardiac surgery is historically based on large doses of intravenous opioids. However, this practice is rapidly changing due to "Enhanced Recovery After Surgery (ERAS)" protocols with proven benefits on morbidity and mortality. Also, the opioid crisis caused by opioid abuse, has changed anaesthesia practice to reduce the use of opioids after surgery. Therefore, perioperative multimodal pain management with regional anaesthesia in minimal invasive cardiac surgery (MICS) has gained a lot of interest.

Serratus Anterior Plane Block (SAPB) is one example of the fascial plane chest wall blocks and aims at achieving complete sensory loss of the anterolateral hemithorax via blockade of the lateral cutaneous branches of the thoracic intercostal nerves (T2-T12). SAPB has already proved its efficacy in thoracic surgery as it reduced pain scores and opioid consumption compared to systemic analgesia in the first 12-24h after surgery. However only few studies investigated the effects of SAPB in minimal invasive cardiac surgery.

Therefore the primary aim of this study is to investigate the analgesic effects of a superficial SAPB in Minimal Invasive Cardiac Surgery compared to a control group with standard intravenous opioid analgesia.

DETAILED DESCRIPTION:
2 x 40 patients scheduled for mitral valve surgery via port access, aortic valve replacement via right anterior thoracotomy and minimal invasive direct coronary artery bypass (MIDCAB) surgery will be randomized in a control or SAPB group.

Every patient will receive the standard anaesthetic treatment. At the end of the surgery, patients in the SAPB group will receive levobupivacaine 0.25 %, 2.5 mg/ml (dosage scheme: 1.25 mg/kg levobupivacaine 0.25%, with a maximum of 100 mg). Levobupivacaine will be given via ultrasound-guided infiltration, in plane, midaxillary, 4-5th rib, between the latissimus dorsi and serratus anterior muscle, at the end of the surgery.

For both the SAPB group and the control group, the ICU nurse will repeatedly administer piritramide 2 mg intravenously, till numerical rating scale (NRS) are less than 4. Also paracetamol 1 g will be continued 4 times daily.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for mitral valve surgery via port access, aortic valve replacement via right anterior thoracotomy and minimal invasive direct coronary artery bypass

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* BMI >35
* Opioid abuse
* Patients known with chronic pain
* Patients known with allergy to local anaesthetics (in this case levobupivacaine)
* Patients known with hypersensitivity to piritramide
* Patients who receive medication that could possibly interact with levobupivacaine (sa. mexiletine, ketoconazole, theophylline)
* Patients who simultaneously participate in another interventional clinical trial, unless the Principal Investigators of the clinical trials give consent by mutual agreement that the patient can participate in another interventional clinical trial
* Soft tissue infection in the area of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Analgesic effect of superficial SAPB in MICS | In the first 48 hours after surgery
  Numeric (pain) Rating Scale every 2 hours
Analgesic effect of superficial SAPB in MICS | In the first 48 hours after surgery
  Total opioid consumption in the intensive care unit

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) | In the first 48 hours after surgery
  PONV every 2 hours
Time to extubation in the intensive care unit | From arrival on the ICU until discharge on the ICU
ICU length of stay | From arrival on the ICU until discharge on the ICU
PaCO2 | In the first 48 hours after surgery
  PaCO2 every 4 hours, calculated by an arterial blood gas test

CONTACTS AND LOCATIONS:
Overall Officials: Steffi Ryckaert, MSc, Study Director — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No